CLINICAL TRIAL: NCT06346600
Title: A Prospective, Non-interventional, Multicenter, Long-term Follow-up Study to Evaluate SKG0106 in the Treatment of Patients With Neovascular (Wet) Age-related Macular Degeneration (nAMD)
Brief Title: A Long-term Follow-up Study to Evaluate SKG0106 in the Treatment of Patients With nAMD
Status: Recruiting | Type: Observational
Sponsor: Skyline Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: SKG0106-LF
Record Dates: First submitted 2024-03-27; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Neovascular (Wet) Age-related Macular Degeneration
Keywords: nAMD; wAMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Long-term Follow-Up of Participants exposed to SKG0106 Dose level 1: No investigational product will be administered in this study.
  Interventions: Genetic: SKG0106
- Long-term Follow-Up of Participants exposed to SKG0106 Dose level 2: No investigational product will be administered in this study.
  Interventions: Genetic: SKG0106
- Long-term Follow-Up of Participants exposed to SKG0106 Dose level 3: No investigational product will be administered in this study.
  Interventions: Genetic: SKG0106

INTERVENTIONS:
Genetic: SKG0106 — Non-interventional (observational) study, long-term follow-up safety and efficacy assessments up to 5 years post SKG0106 injection.

SUMMARY:
This is a Prospective, Non-interventional, Multicenter, Long-term Follow-up Study to Evaluate SKG0106 in the Treatment of Patients with Neovascular (Wet) Age-related Macular Degeneration (nAMD). All subject who completed the parent clinical study (NCT06213038 and NCT05986864) will undergo safety and efficacy assessments up to 5 years post study drug injection.

ELIGIBILITY:
Inclusion Criteria:

Subjects who only meet all of the following criteria are eligible for this study:

* nAMD subjects who have been enrolled in the SKG0106-related study and received SKG0106 injection;
* Subjects who voluntarily sign an informed consent form (ICF) and comply with the protocol to complete the study

Exclusion Criteria:

* Subjects who are judged by the investigator unsuitable for this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is expected that a total of 83 study subjects from parent study will be enrolled. Subjects who meet all the inclusion criteria and for whom none of the exclusion criteria apply will be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Type, severity, and incidence of ocular and systemic adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESIs) | 5 years post study drug injection

SECONDARY OUTCOMES:
Mean change in best corrected visual acuity (BCVA) at each visit from baseline | 5 years post study drug injection
  BCVA of the study eye is examined by the Early Treatment of Diabetic Retinopathy Study (ETDRS) testing at each visit.
Mean change in macular central subfield thickness (CST) at each visit from baseline | 5 years post study drug injection
  Spectral domain optical coherence tomography (SD-OCT) will be performed to measure CST at each visit.
Mean change in patient-reported outcome (VFQ-25) scale scores at each visit from baseline | 5 years post study drug injection
  Both the total scale and subscale scores of the VFQ-25 is ranging from 0 to 100, and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (3):
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Consultants of Texas, Katy, Texas
  - Wagner Macula & Retina Center, Norfolk, Virginia
- China (7):
  - The Second Hospital Of Anhui Medical University, Hefei, Anhui
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Eye Hospital, WMU (Zhejiang Eye Hospital), Wenzhou, Zhejiang
  - Beijing Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - EYE & ENT Hospital of Fudan University, Shanghai
  - Xinhua Hospital Affiliated To Shanghai Jiao Tong University School Of Medicine, Shanghai